CLINICAL TRIAL: NCT05498311
Title: Cosmetic Outcomes Following Conservative Surgery (With or Without Oncoplastic Surgery) for Breast Cancer With Intraoperative Radiotherapy (INTRABEAM) Followed by Hypofractionated External Beam Radiotherapy: a Phase II Trial
Brief Title: Breast Cancer With Intraoperative Radiotherapy Followed by Hypofractionated External Beam Radiotherapy
Acronym: IORT_BREAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IORT BREAST CANCER
Record Dates: First submitted 2021-04-08; First posted 2022-08-12 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Intraoperative radiotherapy; hypofractionated radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Intraoperative Radiotherapy (IORT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Radiotherapy (IORT) (Experimental): Patients with diagnosis of invasive breast cancer (IBC) will be treated with conservative surgery (with or without oncoplastic surgery) and 20 Gy IORT followed by hypofractionated radiotherapy.
  Interventions: Radiation: Intraoperative Radiotherapy (IORT); Procedure: Breast conservative surgery; Radiation: External Beam Hypofractionated Radiotherapy (EBRT)

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy (IORT) — The Intrabeam Photon Radiosurgery System will deliver 20 Gy in the act of breast surgery
Procedure: Breast conservative surgery — Breast conservative surgery with the aim of resecting breast tumour and with or without oncoplastic surgery
Radiation: External Beam Hypofractionated Radiotherapy (EBRT) — A External Beam Hypofractionated Radiotherapy will be administered after surgery. y. The dose per fraction will be 2.67 Gy per session. EBRT will be performed daily from Monday to Friday for fifteen fractions.

SUMMARY:
To evaluate cosmetic outcomes after conservative surgery for breast cancer with INTRABEAM followed by hypofractionated external beam radiotherapy

DETAILED DESCRIPTION:
To evaluate cosmetic outcomes following conservative surgery (with or without oncoplastic surgery) for breast cancer with intraoperative radiotherapy (INTRABEAM) followed by hypofractionated external beam radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of invasive breast carcinoma and eligibility for conservative surgery (with or without oncoplastic surgery) and radiotherapy.
* Not pregnant at diagnosis.
* Signed informed consent form.
* Age ≥45 years old.
* Patients candidates to Intrabeam.
* Patients with ≥60 years with the presence of one or more of the following adverse criteria after surgery:
* Tumor size > 2.5 cm.
* Extensive intraductal carcinoma (≥25%)
* Lymphovascular invasion.
* Involved focal margins (<2mm) without ampliation surgery.

Exclusion Criteria:

* Presence of distant metastasis.
* Primary chemotherapy.
* Lymph node involvement.
* Negative hormonal receptors.
* Diagnosis of any other infiltrating tumour except for adequately resected squamous or basal cell epitheliomas
* Patients with collagen vascular disease (systemic lupus erythematosus, scleroderma, dermatomyositis).
* Uncontrolled infection.
* Concurrent treatment with other experimental treatments
* Lack of signed informed consent form.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2016-10-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Cosmetic results - BCCT | Baseline and every 12 months until 60 months
  It will be measured by the BCCT.core software programme. This software uses 4 photographies of the breast for each timepoint and evaluates cosmetic outcome based upon symmetry, skin colour changes and surgical scar appearance. The lower the calculated score, the better the cosmetic outcome (1=excellent, 2=good, 3=fair, 4=poor)
Changes in Cosmetic results - Self Evaluation using YBT | Baseline and every 12 months until 60 months
  Questionnaire for cosmetic self-evaluation from the Young Boost Trial (YBT) that consists s of 8 questions about various aspects (size, shape, skin colour, massiveness of the breast, nipple position, general appearance, visibility of the surgical scar, and overall satisfaction) to evaluate the degree of satisfaction of the patients themselves about the cosmetic results.

SECONDARY OUTCOMES:
Changes in Quality of life (QOL) - General | Baseline and every 12 months until 60 months
  It will be measured by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaires QLQ-C30
Toxicity (acute and late) | Baseline and every 12 months until 60 months
  Defined according to the NCI criteria published in the Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Local control | Baseline and every 3 months after completion of EBRT and thereafter every 6 months for 5 years
  Defined as histologically-confirmed evidence of tumour recurrence in the ipsilateral breast
Changes in Quality of life (QOL) - Breast | Baseline and every 12 months until 60 months
  It will be measured by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaires QLQ-BR23

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Martínez, MD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Evelyn Martínez, L'Hospitalet de Llobregat, Barcelona, Spain